CLINICAL TRIAL: NCT06092697
Title: Evaluation of 3D Printed Polyether Ether Ketone (PEEK) and Milled PEEK Indirect Restorations Compared to Hybird Resin Composite Indirect Restorations Over One Year Period of Time ( A Randomized Clinical Trial )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Ahmed Abdalnaby Ahmed Attia, Lecturer Assistant at MSA UNIVERSITY, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Hadeer'sPROTOCOL-PHD
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Clinical Performance

STUDY DESIGN:
Intervention Model Description: A superiority frame randomized, controlled, parallel clinical trial with 1:1 allocation ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3D printed PEEK (Experimental): Indirect dental restoration
  Interventions: Other: 3D printed PEEK restorations
- Milled PEEK (Experimental): Indirect dental restoration
  Interventions: Other: 3D printed PEEK restorations
- Hybird resin composite (Active Comparator): Indirect dental restoration
  Interventions: Other: 3D printed PEEK restorations

INTERVENTIONS:
Other: 3D printed PEEK restorations — Indirect dental restoration
  Other Names: Milled PEEK

SUMMARY:
Clinical performance evaluation of 3D Printed Polyether ether ketone (PEEK) and milled PEEK indirect restorations compared to hybird resin composite indirect restorations over one year period of time

DETAILED DESCRIPTION:
The aim of this study is to evaluate fracture and retention, wear of 3D printed PEEK indirect restorations and milled PEEK indirect restorations compared to milled indirect hybrid resin composite restorations according to FDI criteria over one year.

According to indirect restorations cavity preparation principles, shade selection and occlusal examination will be done preoperatively, followed by cavity preparations that will be carried out with tapered diamond stones.

The prepared teeth for the indirect restorations will be scanned with an optical scanner. Then restorations will be designed by a CAD software and files will be made in STL format, so as to be ready for either 3D printing or milling with different materials.

While the printed PEEK restorations are additively made, the milled PEEK and hybrid composite restorations are both milled out of either a disc or block ( size 12) using a CAD/CAM milling machine.

After the printing and the milling procedures are complete, the restorations are then promptly removed. Each restoration will be assessed and adjusted for its cavity after the occlusal surface is recontoured. This post-processing adjustments will be applied to both 3d printed ones and milled restorations. After assessment and needed adjustments are done, all restorations will be cemented into the cavities in accordance with the manufacturer's recommendations.

For each recall examination, two independent evaluators will perform the direct clinical evaluation for the fracture and retention at baseline, after 6 and 12 months using written criteria based on FDI world dental federation criteria. Together with the wear testing that will be performed by scanning of the restoration surfaces at baseline, after 6 and 12 months. Using parallel confocal technology, a 3D dental scanner (CEREC Primescan; Sirona, Bensheim, Germany) to attain the 3D Standard Tessellation Language (STL) models will be used. These scan models will be then introduced through a wear measuring software (Geomagic Design X; 3D Systems, Seoul, Korea) which will import, analyze, and superimpose the digitalized 3D models. So, it will automatically calculate the amount of occlusal volume lose due to wear.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging (18-45) years.
* Patients with a high level of oral hygiene.
* Each patient enrolled in the study should have moderate carious lesion or defective restoration needs to be replaced on a mandibular permanent molar.
* Patients with ability to attend periodical follow-ups.

Exclusion Criteria:

* Patients with general/systemic diseases or allergies.
* Patients with chronic use of anti- inflammatory, analgesic, and psychotropic drugs.
* Pregnant or lactating females.
* Patients with parafunctional habits.
* Patients with experience of allergic reactions against any components of the used materials.
* Patients receiving orthodontic treatment.
* Inability to comply with study procedures.
* Collateral participation in another research study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Fracture and retention (Category F1)(Revised FDI criteria for evaluating direct and indirect dental restorations- recommendations for its clinical use, interpretation, and reporting) | Baseline, 6 months, 12 months
  Outcome:Fracture of the material and retention Measuring device: Revised FDI criteria for evaluating direct and indirect dental restorations- recommendations for its clinical use, interpretation, and reporting.
  (Hickel et al., 2023) Measuring unit: Scoring system (Ordinal) 1. Clinically excellent/very good (sufficient) 2. Clinically good (sufficient) 3. Clinically satisfactory (sufficient) 4. Clinically unsatisfactory (partially insufficient) 5. Clinically poor (entirely insufficient)

SECONDARY OUTCOMES:
occlusion and wear (Category F5) | Baseline, 6 months, 12 months
  Wear potential of the restoration Measuring device: A. Digital scanner (CEREC Primescan intraoral Scanner) B. Geometrical Subtraction software (Geomagic control software) (Tang et al. 2021) Measuring unit : Microns (Quantitative)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abhay SS, Ganapathy D, Veeraiyan DN, Ariga P, Heboyan A, Amornvit P, Rokaya D, Srimaneepong V. Wear Resistance, Color Stability and Displacement Resistance of Milled PEEK Crowns Compared to Zirconia Crowns under Stimulated Chewing and High-Performance Aging. Polymers (Basel). 2021 Oct 30;13(21):3761. doi: 10.3390/polym13213761. PMID 34771318